CLINICAL TRIAL: NCT02619071
Title: ChEmo-Genomics Based Treatment of Acute Myeloid Leukemia- CeGAL-IPC 2014-012
Brief Title: ChEmo-Genomics Based Treatment of Acute Myeloid Leukemia
Acronym: CeGAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Cancer Research Center of Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CeGAL-IPC-2014-012
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: acute myeloid leukemia- refractory AML- relapsed AML- precision medecine-
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refractory or relapsed acute myeloid leukemia (Experimental)
  Interventions: Procedure: Tumor sampling; Biological: Constiutional DNA sampling

INTERVENTIONS:
Procedure: Tumor sampling — Bone marrow aspirate, blood sampling
Biological: Constiutional DNA sampling — Buccal swab or Hair follicles

SUMMARY:
Adult acute myeloid leukemia (AML) is a heterogeneous hematologic malignancy associated with poor prognosis, especially after relapse. High-throughput genomic studies have highlighted the importance of molecular alteration in the pathophysiology, clinical evolution and treatment response of AML. In addition, identification of specific gene mutation can be targeted by specific inhibitors, opening the way to personalized treatments. However, only a limited number of gene mutations are druggable or actionable, highlighting the need for additional information to guide treatment choices. Among them, new Drug Screening Tests (DST) allow for the screening of library of hundreds of drugs to ex-vivo patient-derived AML cells. Combination of genomic and pharmacologic approaches might therefore improve prediction of drug effects. There is an urgent need to bring these approaches into the clinic but feasibility trials are necessary before incorporating them into treatments strategies.The proposed study is a prospective multicentre feasibility study of a combined "chemo-genomic" approach in patients with advanced AML.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of acute myeloid leukemia according to WHO classification
* Refractory or relapsed disease
* ECOG performance status of <3
* Life expectancy >3 months
* Written informed consent
* Affiliation to the French Social Security System.

Exclusion Criteria:

* Diagnosis of Acute Promyelocytic Leukemia.
* Patients deprived of liberty or placed under the authority of a tutor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients for whom a treatment tailored according to chemogenomic data could be proposed to the investigator within a 21 days time-frame in at least 30% of cases. | 24 months

SECONDARY OUTCOMES:
Correlations between genomic alterations (identified by mutatome and transcriptome analyses) and drug sensitivity profiles | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut PAOLI-CALMETTES, Marseille, France

REFERENCES:
- [Derived] Collignon A, Hospital MA, Montersino C, Courtier F, Charbonnier A, Saillard C, D'Incan E, Mohty B, Guille A, Adelaide J, Carbuccia N, Garnier S, Mozziconacci MJ, Zemmour C, Pakradouni J, Restouin A, Castellano R, Chaffanet M, Birnbaum D, Collette Y, Vey N. A chemogenomic approach to identify personalized therapy for patients with relapse or refractory acute myeloid leukemia: results of a prospective feasibility study. Blood Cancer J. 2020 Jun 3;10(6):64. doi: 10.1038/s41408-020-0330-5. PMID 32488055